CLINICAL TRIAL: NCT04337580
Title: A Phase II Trial of FASN Inhibition by Omeprazole in Combination With Cabazitaxel in Patients With Docetaxel- and Castration-Resistant Prostate Cancer
Brief Title: Fatty Acid Synthase Inhibition in Castration Refractory Prostate Cancer
Acronym: FASN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00068039; P30CA012197 (NIH); WFBCC 85220 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2020-04-02; First posted 2020-04-07 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer; Refractory Cancer; Castration Resistant Prostatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Prostatic Neoplasms, Castration-Resistant | interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Omeprazole Plus Standard of Care for Prostate Cancer Regimen (Experimental): This intervention will be given on an outpatient basis. Omeprazole, 80 mg twice daily.
  Interventions: Drug: Omeprazole 80 mg twice daily

INTERVENTIONS:
Drug: Omeprazole 80 mg twice daily — Participants will be treated with omeprazole 80 mg twice daily on Day 0. Within 10 days of starting omeprazole, participants will be treated with standard prostate cancer dosing of every three week docetaxel or cabazitaxel based on package insert. Participants that have only had docetaxel will be retreated with docetaxel along with concurrent omeprazole. Patients that have had both docetaxel and cabazitaxel will be retreated with either cabazitaxel or docetaxel (investigators choice) along with concurrent omeprazole. However investigators encourage investigator to choose cabazitaxel in patients previously treated with cabazitaxel.

SUMMARY:
The purpose of this research study is to find out what effects (good and bad) omeprazole and cabazitaxel, or omeprazole and docetaxel, has on participants and their condition. Investigators believe omeprazole may help the other medications work.

DETAILED DESCRIPTION:
Primary Objective(s): Obtain Overall Response Rate (ORR) to taxane therapy by adding the fatty acid synthase inhibitor, omeprazole to the current "failing" taxane regimen in 15% of subjects using Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria, defined by partial response (PR) or complete response (CR)

Secondary Objectives (only at patients treated at Wake Forest Baptist Comprehensive Cancer Center main campus):

* Pharmacodynamics-demonstrate omeprazole in vivo fatty acid synthase inhibition by 11C-Acetate PET/CT (3-6) Non-invasive approach to demonstrate the fatty acid synthase inhibitor (omeprazole) is hitting its target
* Obtain a prostate specific antigen response rate by adding the fatty acid synthase inhibitor omeprazole to the current "failing" taxane regimen. (16)
* Measure pain using the Patient-Reported Outcomes Measurement Information System (PROMIS) at Baseline, Cycle 5, Cycle 12, and every cycle thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have castrate refractory prostate cancer with prior taxane treatment (docetaxel or cabazitaxel) which was used in the castrate refractory setting
* Cancer Progression as defined by PCWG3
* Age 18 or older.
* ECOG 0, 1, or 2
* Life expectancy of greater than 2 months
* Men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).
* Organ & marrow function as defined below: Absolute neutrophil count >1,200/mcL Platelets >75,000/mcL; total bilirubin= within normal institutional limits; AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal; creatinine <2.5 X institutional upper limit of normal

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to omeprazole or taxane therapy.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Change Radiographic Response - RECIST 1.1 | At 3, 6 and 9 months
  Response will be defined by RECIST 1.1 as defined by Prostate Cancer Clinical Trials Working Group 3 definition for complete response (CR) - disappearance of all target lesions); partial response (PR) (at least a 30% decrease in the sum of diameters of target lesions); progressive disease (PD) (at least a 20% increase in the sum of diameters or target lesions); stable disease (SD) (neither sufficient shrinkage to qualify for partial response nor sufficient to qualify for progressive disease); or not evaluable (NE).
Change in Bone Metastasis Response - Prostate Cancer Clinical Trials Working Group 3 (PCWG3) | At 3, 6 and 9 months
  Response will be defined by Prostate Cancer Clinical Trials Working Group 3 (PCWG3) for complete response (CR), partial response (PR), progressive disease (PD), stable disease (SD) or not evaluable (NE).

SECONDARY OUTCOMES:
Fatty Acid Synthase Activity - Pre Omeprazole Use | At baseline
  Performed only on the first 10 participants by utilizing the 11C acetate tracer in the PET scan to evaluate the fatty acid synthase activity prior to omeprazole by examining changes in the values of standardized uptake. we will perform a two-sample t-test to see whether the change in SUV values is different between patients with an objective response versus those without an objective response.
Fatty Acid Synthase Activity - Post Omeprazole Use | Up to approximately 2 years
  Evaluating the first 10 participants by utilizing the 11C acetate tracer in the PET scan to evaluate the fatty acid synthase activity prior to omeprazole by examining changes in the values of standardized uptake. we will perform a two-sample t-test to see whether the change in SUV values is different between patients with an objective response versus those without an objective response.
Prostate Specific Antigen (PSA) Progression | At baseline and up to approximately 2 years
  Investigators will collect PSA to determine whether PSA progression is positive or negative. Positive meaning that PSA slope is getting worse over time than it was prior to treatment and negative meaning PSA slope is improving after treatment when compared to baseline.
Prostate Specific Antigen (PSA) Response | At baseline and up to approximately 2 years
  Investigators will examine a PSA response rate (baseline on clinical definition of PSA response). In this analysis investigators will determine for each participant if they are a PSA responder (yes/no) and then using this data will estimate a 95% exact Clopper Pearson binomial interval for the PSA response rate.
Patient Reported Outcome - Pain | At baseline, 12 weeks, and Day 1 of every subsequent cycle (each cycle is 28 days) up to approximately 2 years
  Participants will report pain intensity at Cycle 1 Day 1 (baseline) compared to Cycle 5, Day 1 and Day 1 of every subsequent cycle on numeric scale of 0-to-10 (0 = no pain, 10 = worse imaginable pain). A paired t-test will be performed to determine whether the Pain score improved or worsened in patients after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goodman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - W.G. Bill Hefner VA Medical Center, Salisbury, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No